CLINICAL TRIAL: NCT01737268
Title: Long-term Study of FK949E in Elderly Patients -Long-term Study in Elderly Bipolar Disorder Patients With Major Depressive Episodes-
Brief Title: Long-term Study of FK949E in Elderly Bipolar Disorder Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6949-CL-0022
Record Dates: First submitted 2012-11-08; First posted 2012-11-29 (Estimated); Results first posted 2017-10-31 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-10

CONDITIONS: Bipolar Disorder; Elderly
Keywords: patients; Major depressive episode; FK949E
MeSH Terms: conditions — Bipolar Disorder | interventions — Quetiapine Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FK949E Elderly Participants (Experimental): After 2 days of dose-titration, elderly participants received either FK949E 150 mg or FK949E 300 mg once daily at bedtime from day 3 to week 52. Dose increase and reduction was allowed following dose increase or reduction guidelines and at the investigator's discretion. After which, participants went through a follow-up period of 1 week. For participants, who completed or discontinued treatment at FK949E 300 mg, a dose-tapering period was placed before proceeding to the follow-up period, and FK949E 150 mg was administered once daily for 1 week in this period.
  Interventions: Drug: FK949E

INTERVENTIONS:
Drug: FK949E — Oral tablet
  Other Names: quetiapine

SUMMARY:
FK949E was administered to elderly bipolar disorder patients with major depressive episode for 52 weeks. Its safety, efficacy, and plasma concentration change were evaluated in an open-label manner.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bipolar I or II disorder as specified in the Diagnostic and Statistical Manual of Mental Disorders, 4th edition, Text Revision (DSM-IV-TR), with a major depressive episode
* Able to participate in the study with understanding of and compliance with subject requirements during the study in the investigator's or subinvestigator's opinion
* Male subjects must agree to take appropriate contraceptive measures with condoms during the study period.
* Female subjects must be confirmed to have no childbearing potential during the study period

Exclusion Criteria:

* Concurrent or previous history of DSM-IV-TR Axis I disorders, except bipolar disorder, within the last 6 months before informed consent
* Concurrence of DSM-IV-TR Axis II disorder that was considered to greatly affect patient's current mental status.
* The Young Mania Rating Scale (YMRS) total score of 13 points or more.
* Nine or more mood episodes within the last 12 months before informed consent.
* Lack of response to at least 6-week treatment with at least 2 antidepressants for the current major depressive episode in the investigator's or subinvestigator's opinion
* The current major depressive episode persisting for more than 12 months or less than 4 weeks before informed consent.
* History of substance dependence (other than caffeine and nicotine) or alcohol abuse or dependence.
* Treatment with a depot antipsychotic within the last 49 days before primary registration.
* Unable to suspend antipsychotics or antidepressants after primary registration
* Treatment with two or more of mood stabilizers (lithium carbonate and/or sodium valproate) and lamotrigine, if these drugs, except one of either drug, cannot be suspended after primary registration.
* Unable to suspend antiepileptics (except lamotrigine and sodium valproate), antianxiety agents, hypnotics, sedatives, psychostimulants, antiparkinsonian agents, cerebral ameliorators, antidementia agents, or anorectics, except those specified as conditionally-allowed concomitant drugs, from 7 days before primary registration
* Electroconvulsive therapy within the last 83 days before primary registration.
* A possible need of psychotherapy during the study period (unless the therapy has been commenced at least 83 days before primary registration).
* The Hamilton Depression Rating Scale (HAM-D17) suicide score of 3 points or more, history of suicide attempt within the last 6 months before informed consent, or the risk of suicide in the investigator's or subinvestigator's opinion

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-10-29 (Actual); Primary Completion 2016-06-29 (Actual); Study Completion 2016-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (32):
- Japan (32):
  - Site JP00024, Chiba
  - Site JP00023, Fukuoka
  - Site JP00025, Fukuoka
  - Site JP00015, Fukushima
  - Site JP00029, Fukushima
  - Site JP00001, Hokkaido
  - Site JP00002, Hokkaido
  - Site JP00003, Hokkaido
  - Site JP00004, Hokkaido
  - Site JP00005, Hokkaido
  - Site JP00006, Hokkaido
  - Site JP00007, Hokkaido
  - Site JP00008, Hokkaido
  - Site JP00009, Hokkaido
  - Site JP00010, Hokkaido
  - Site JP00011, Hokkaido
  - Site JP00012, Hokkaido
  - Site JP00013, Hokkaido
  - Site JP00028, Hyōgo
  - Site JP00031, Ibaraki
  - Site JP00017, Kanagawa
  - Site JP00032, Kanagawa
  - Site JP00019, Kumamoto
  - Site JP00018, Kyoto
  - Site JP00014, Osaka
  - Site JP00016, Tokyo
  - Site JP00020, Tokyo
  - Site JP00021, Tokyo
  - Site JP00022, Tokyo
  - Site JP00026, Tokyo
  - Site JP00027, Tokyo
  - Site JP00030, Tottori

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Fukushi R, Nomura Y, Katashima M, Komatsu K, Sato Y, Takada A. Approach to Evaluating QT Prolongation of Quetiapine Fumarate in Late Stage of Clinical Development Using Concentration-QTc Modeling and Simulation in Japanese Patients With Bipolar Disorder. Clin Ther. 2020 Aug;42(8):1483-1493.e1. doi: 10.1016/j.clinthera.2020.06.002. Epub 2020 Aug 11. PMID 32792252
- See also: Link to results on Astellas Clinical Study Results website — https://www.astellasclinicalstudyresults.com/study.aspx?ID=214

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Elderly participants with documented clinical diagnosis meeting the Diagnostic and Statistical Manual of Mental Disorders, 4th edition, Text Revision criteria for bipolar I disorder or bipolar II disorder, with most recent episode depressed confirmed by the Mini-International Neuropsychiatric Interview were recruited from 32 sites in Japan.
Pre-assignment Details: Participants who were not taking quetiapine or was at < 50 mg/day at least 28 days prior to informed consent, FK949E was administered at an initial dose of 50 mg during the dose-titration period. Participants who were taking quetiapine at 50 to < 300 mg/day or 300 mg/day, FK949E was administered at 150 mg/day during the dose-titration period.
Period: Overall Study
Arm/Group | FK949E Elderly Participants
Started | 20
Treated | 20
Completed | 11
Not Completed | 9
Not completed — Adverse Event | 6
Not completed — Worsening of Target Disease | 2
Not completed — In consideration of the patient's safety | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS), which consisted of participants who received at least one dose of the study drug and were evaluated for at least one efficacy variable after the start of treatment with the study drug.
Arm/Group | FK949E Elderly Participants
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.9 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 8
Montgomery-Asberg Depression Rating Scale (MADRS) Total Score [Mean (Standard Deviation); unit: Units of a scale] — The MADRS is a 10-item scale to measure the severity of depressive episodes, where each item is rated on a scale from 0 to 6. The MADRS total score ranges from 0 to 60 with lower scores indicating less depressive symptoms. Population: FAS
  Units of a scale | 25.1 (6.4)
Hamilton Depression Scale (HAM-D17) Total Score [Mean (Standard Deviation); unit: Units of a scale] — The HAM-D17 is a clinician-rated 17-item scale for assessing the severity of depression symptoms. The scores for each item range from 0 to 4 or 0 to 2, where 0 represents no symptoms. The rating is based on the past 7 days prior to the time of assessment. The total score ranges from 0 to 52 with lower scores indicating less depressive symptoms. Population: FAS
  Units of a scale | 19.3 (4.9)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Last Assessment in Treatment Period in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score
Description: The MADRS is a 10-item scale to measure the severity of depressive episodes, where each item is rated on a scale from 0 to 6. The MADRS total score ranges from 0 to 60 with lower scores indicating less depressive symptoms.
Time Frame: Baseline and week 52 (or the time of last assessment for participants who discontinued earlier)
Population: FAS population; last assessment value is used for participants who discontinued before week 52.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FK949E Elderly Participants
Number analyzed (Participants) | 19
units on a scale | -13.1 (11.0)

2. Secondary Outcome: Change From Baseline to Last Assessment in Treatment Period in Hamilton Depression Scale (HAM-D17)
Description: The HAM-D17 is a clinician-rated 17-item scale for assessing the severity of depression symptoms. The scores for each item range from 0 to 4 or 0 to 2, where 0 represents no symptoms. The rating is based on the past 7 days prior to the time of assessment. The total score ranges from 0 to 52 with lower scores indicating less depressive symptoms.
Time Frame: Baseline and week 52 (or the time of last assessment for participants who discontinued earlier)
Population: FAS population; last assessment value is used for participants who discontinued before week 52.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FK949E Elderly Participants
Number analyzed (Participants) | 19
units on a scale | -10.5 (8.2)

3. Secondary Outcome: Change From Baseline to Last Assessment in Treatment Period in Clinical Global Impression-Bipolar-Severity of Illness (CGI-BP-S): Overall Bipolar Illness
Description: The CGI-BP-S is a scale which assesses a participant's severity of their overall bipolar illness, depression, and mania as assessed by the clinician using a scale from with the scale from 1 (Normal, not ill) to 7 (very severely ill).
Time Frame: Baseline and week 52 (or the time of last assessment for participants who discontinued earlier)
Population: FAS population; last assessment value is used for participants who discontinued before week 52.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FK949E Elderly Participants
Number analyzed (Participants) | 19
units on a scale | -1.2 (1.5)

4. Secondary Outcome: Change From Baseline to Last Assessment in Treatment Period in CGI-BP-S: Depression
Description: as for outcome 3
Time Frame: Baseline and week 52 (or the time of last assessment for participants who discontinued earlier)
Population: FAS population; last assessment value is used for participants who discontinued before week 52.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FK949E Elderly Participants
Number analyzed (Participants) | 19
units on a scale | -1.3 (1.5)

5. Secondary Outcome: Change From Baseline to Last Assessment in Treatment Period in CGI-BP-S: Mania
Description: as for outcome 3
Time Frame: Baseline and and week 52 (or the time of last assessment for participants who discontinued earlier)
Population: FAS population; last assessment value is used for participants who discontinued before week 52.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FK949E Elderly Participants
Number analyzed (Participants) | 19
units on a scale | 0 (0)

6. Secondary Outcome: Clinical Global Impression-Bipolar-Change (CGI-BP-C): Overall Bipolar Illness
Description: The CGI-BP-C is a scale which assesses the degree of change or improvement from baseline for each of overall bipolar illness, depression and mania, by grading it using 8 grades, from 1 (very much improved) to 7 (very much worse) or 8 (not applicable). Grade 8 (not applicable) was regarded as a missing value for purposes of calculating the mean score.
Time Frame: Week 52 (or the time of last assessment for participants who discontinued earlier)
Population: FAS population; last assessment value is used for participants who discontinued before week 52.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FK949E Elderly Participants
Number analyzed (Participants) | 19
units on a scale | 2.4 (1.3)

7. Secondary Outcome: CGI-BP-C: Depression
Description: as for outcome 6
Time Frame: Week 52 (or the time of last assessment for participants who discontinued earlier)
Population: FAS population; last assessment value is used for participants who discontinued before week 52.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- FK949E Elderly Participant: After 2 days of dose-titration, elderly participants received either FK949E 150 mg or FK949E 300 mg once daily at bedtime from day 3 to week 52. Dose increase and reduction was allowed following dose increase or reduction guidelines and at the investigator's discretion. After which, participants went through a follow-up period of 1 week. For participants, who completed or discontinued treatment at FK949E 300 mg, a dose-tapering period was placed before proceeding to the follow-up period, and FK949E 150 mg was administered once daily for 1 week in this period
Arm/Group | FK949E Elderly Participant
Number analyzed (Participants) | 19
units on a scale | 2.4 (1.3)

8. Secondary Outcome: CGI-BP-C: Mania
Description: as for outcome 6
Time Frame: Week 52 (or the time of last assessment for participants who discontinued earlier)
Population: FAS population; last assessment value is used for participants who discontinued before week 52.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FK949E Elderly Participants
Number analyzed (Participants) | 19
units on a scale | 4.0 (0.0)

9. Secondary Outcome: Number of Participants With Adverse Events
Description: An adverse event (AE) is defined as any undesirable or unintended sign (including abnormal laboratory test values), symptom, or disease occurring while the study drug was administered, regardless of whether or not there was a causal relationship with the study drug. A serious AE is defined as a an event resulting in death, persistent or significant disability/incapacity or congenital anomaly or birth defect, was life-threatening, re quire d or prolonged hospitalization or was considered medically important.
Time Frame: From first dose of study drug up to week 52 (52 weeks)
Population: Safely Analysis Set (SAF), which included participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | FK949E Elderly Participants
Number analyzed (Participants) | 20
Participants
  Any AE | 18
  Drug-related AEs | 18
  Deaths | 0
  Serious AEs | 2
  Drug-related SAEs | 1
  AEs that caused study drug discountinuation | 8
  Drug-related AEs that caused study drug discont. | 7

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to week 52 (52 weeks)
Arm/Group | FK949E Elderly Participants
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 2/20
Other Adverse Events (participants affected / at risk) | 18/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FK949E Elderly Participants (N=20)
Malaise (General disorders) | 1
Depression (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FK949E Elderly Participants (N=20)
Hypothyroidism (Endocrine disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Salivary hypersecretion (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Malaise (General disorders) | 3
Thirst (General disorders) | 7
Influenza (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 4
Fall (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 1
Blood creatine phosphokinase increased (Investigations) | 1
Blood glucose decreased (Investigations) | 1
Blood prolactin increased (Investigations) | 4
Blood thyroid stimulating hormone increased (Investigations) | 2
Blood triglycerides increased (Investigations) | 1
Blood uric acid increased (Investigations) | 1
Liver function test abnormal (Investigations) | 1
Weight decreased (Investigations) | 1
Platelet count increased (Investigations) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 4
Dizziness postural (Nervous system disorders) | 1
Dysarthria (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Movement disorder (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 11
Depression (Psychiatric disorders) | 1
Intentional self-injury (Psychiatric disorders) | 1
Rosacea (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1
Gait disturbance (General disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment.